CLINICAL TRIAL: NCT02204618
Title: Cochlear Implantation in Single Sided Deafness and Asymmetrical Hearing Loss: a Cost/Utility Study.
Acronym: CISSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 7053 10; PRME2013 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Retrocochlear Pathology; Auditory Processing Disorder, Central; Major Cochlear Ossification or Malformation
Keywords: single sided deafness; Asymmetrical hearing loss; Cost-utility; Tinnitus; Cochlear implants; Bone conduction device; Dichotic hearing; Squelch effect.
MeSH Terms: conditions — Language Development Disorders; Congenital Abnormalities; Tinnitus | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cochlear implantation (Experimental): Our experimental protocol relies on real life therapeutic strategy, where a cochlear implant may be proposed once CROS and bone conductions systems have failed. Thus, all subjects enrolled in our study will try CROS and bone conduction devices. If these trials are ineffective, the remaining subjects will be randomized between two arms (cochlear implantation vs 6 months abstention followed by cochlear implantation).
  Interventions: Device: cochlear implantation
- 6 months initial abstention (Other): Our experimental protocol relies on real life therapeutic strategy, where a cochlear implant may be proposed once CROS and bone conductions systems have failed. Thus, all subjects enrolled in our study will try CROS and bone conduction devices. If these trials are ineffective, the remaining subjects will be randomized between two arms (cochlear implantation vs 6 months abstention followed by cochlear implantation).
  Interventions: Other: 6 months initial abstention

INTERVENTIONS:
Device: cochlear implantation
  Arms: cochlear implantation
Other: 6 months initial abstention — Our experimental protocol relies on real life therapeutic strategy, where a cochlear implant may be proposed once CROS and bone conductions systems have failed. Thus, all subjects enrolled in our study will try CROS and bone conduction devices. If these trials are ineffective, the remaining subjects will be randomized between two arms (cochlear implantation vs 6 months abstention followed by cochlear implantation).
  Arms: 6 months initial abstention

SUMMARY:
The investigators assume that cochlear implants in this indication are not only effective but also cost-effective. The investigators' experimental protocol relies on real life therapeutic strategy, where a cochlear implant may be proposed once CROS and bone conductions systems have failed. Thus, all subjects enrolled in our study will try CROS and bone conduction devices. If these trials are ineffective, the remaining subjects will be randomized between two arms (cochlear implantation vs 6 months abstention followed by cochlear implantation). A comparative cost-utility analysis between the two arms, of medical consequences measured in terms of quality of life will identify a preference for a strategy. Specific binaural hearing measurements with respect to each treatment option (abstention, CROS, bone conduction device, cochlear implant) will also be collected.

DETAILED DESCRIPTION:
Single sided deafness and profound asymmetrical hearing loss are impairments that significantly alter quality of life. Behavioural problems and scholar delays have been reported in children. Speech recognition with background or competing noise and sound localization are both impaired. 1/1000 new borns are affected and the incidence tends to rise in the adult population. At the moment, there is no guideline regarding the treatment of single sided deafness and asymmetrical hearing loss. Some patients don't even receive any therapeutic proposition.

Three treatment options are available :

* CROS (Contralateral Routing Of the Signal) systems that convey the auditory information from the deaf ear to the good ear using wi-fi
* bone conduction devices which use transcranial conduction to convey auditory information from the poor ear to the good ear
* cochlear implants that directly stimulate afferent fibers of auditory nerve in the poor ear Cochlear implantation is therefore the only treatment which restores stimulation in the poor ear. Its efficacy in single sided deafness associated with incapacitating tinnitus have been demonstrated by Pr Van de Heyning (Leeuven, Be) and colleagues. Its interest has been compared to CROS systems and bone conduction devices in a valuable study conducted by S. Arndt (Pr Laszig, Freibourg, Ger). Cochlear implants provided better speech in noise recognition scores in dichotic hearing, i.e when speech and noise sources are spatially separated. Their first publication involved 11 patients but to date, more than 110 patients with single sided deafness have been included in their protocol. The efficacy of cochlear implantation has thus been validated in the treatment of single sided deafness and asymmetrical hearing loss.

The investigators assume that cochlear implants in this indication are not only effective but also cost-effective. The investigators' experimental protocol relies on real life therapeutic strategy, where a cochlear implant may be proposed once CROS and bone conductions systems have failed. Thus, all subjects enrolled in our study will try CROS and bone conduction devices. If these trials are ineffective, the remaining subjects will be randomized between two arms (cochlear implantation vs 6 months abstention followed by cochlear implantation). A comparative cost-utility analysis between the two arms, of medical consequences measured in terms of quality of life will identify a preference for a strategy. Specific binaural hearing measurements with respect to each treatment option (abstention, CROS, bone conduction device, cochlear implant) will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Single sided deafness or profound asymmetrical hearing loss confirmed using pure tone audiometry and auditory brainstem responses, with or without tinnitus
* Written consent to the protocol

Exclusion Criteria:

* Retrocochlear pathology (vestibular schwannoma, severe central auditory processing disorder)
* Major cochlear ossification or malformation
* Subjects under juridical protections or tutelage measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
incremental cost-utility ratio | 6 months after cochlear implantation versus no treatment option

SECONDARY OUTCOMES:
Global score of EuroQoL-5D | before and after auditory rehabilitation (cochlear implantation, CROS system or bone conduction device): Day 0, Week 3, Week 6, Month 6
Global score of Nijmegen Cochlear implant Questionnaire (NCIQ) | before and after auditory rehabilitation (cochlear implantation, CROS system or bone conduction device): Day 0, Week 3, Week 6, Month 6
Nijmegen Cochlear Implant Questionnaire (NCIQ): score in advanced auditory perception section | before and after auditory rehabilitation (cochlear implantation, CROS system or bone conduction device): Day 0, Week 3, Week 6, Month 6
Speech Reception Thresholds | before and after auditory rehabilitation (cochlear implantation, CROS system or bone conduction device): Day 0, Week 3, Week 6, Month 6
  Signal to noise ratio that allows 50% words recognition) in diotic hearing, dichotic hearing and reverse dichotic hearing
Mean error angle for sound localization | before and after auditory rehabilitation (cochlear implantation, CROS system or bone conduction device): Day 0, Week 3, Week 6, Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse - Pierre Paul Riquet Hospital, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Van de Heyning P, Vermeire K, Diebl M, Nopp P, Anderson I, De Ridder D. Incapacitating unilateral tinnitus in single-sided deafness treated by cochlear implantation. Ann Otol Rhinol Laryngol. 2008 Sep;117(9):645-52. doi: 10.1177/000348940811700903. PMID 18834065
- [Background] Plontke SK, Heider C, Koesling S, Hess S, Bieseke L, Goetze G, Rahne T. Cochlear implantation in a child with posttraumatic single-sided deafness. Eur Arch Otorhinolaryngol. 2013 May;270(5):1757-61. doi: 10.1007/s00405-013-2350-2. Epub 2013 Jan 29. PMID 23358584
- [Background] Vermeire K, Van de Heyning P. Binaural hearing after cochlear implantation in subjects with unilateral sensorineural deafness and tinnitus. Audiol Neurootol. 2009;14(3):163-71. doi: 10.1159/000171478. Epub 2008 Nov 13. PMID 19005250
- [Background] Punte AK, Vermeire K, Hofkens A, De Bodt M, De Ridder D, Van de Heyning P. Cochlear implantation as a durable tinnitus treatment in single-sided deafness. Cochlear Implants Int. 2011 May;12 Suppl 1:S26-9. doi: 10.1179/146701011X13001035752336. PMID 21756468
- [Background] Lazard DS, Marozeau J, McDermott HJ. The sound sensation of apical electric stimulation in cochlear implant recipients with contralateral residual hearing. PLoS One. 2012;7(6):e38687. doi: 10.1371/journal.pone.0038687. Epub 2012 Jun 19. PMID 22723876
- [Background] Persson P, Harder H, Arlinger S, Magnuson B. Speech recognition in background noise: monaural versus binaural listening conditions in normal-hearing patients. Otol Neurotol. 2001 Sep;22(5):625-30. doi: 10.1097/00129492-200109000-00011. PMID 11568669
- [Background] Bess FH. The minimally hearing-impaired child. Ear Hear. 1985 Jan-Feb;6(1):43-7. doi: 10.1097/00003446-198501000-00012. PMID 4038669
- [Background] Bovo R, Martini A, Agnoletto M, Beghi A, Carmignoto D, Milani M, Zangaglia AM. Auditory and academic performance of children with unilateral hearing loss. Scand Audiol Suppl. 1988;30:71-4. PMID 3227285
- [Background] Lieu JE. Speech-language and educational consequences of unilateral hearing loss in children. Arch Otolaryngol Head Neck Surg. 2004 May;130(5):524-30. doi: 10.1001/archotol.130.5.524. PMID 15148171
- [Background] Giolas TG, Wark DJ. Communication problems associated with unilateral hearing loss. J Speech Hear Disord. 1967 Nov;32(4):336-43. doi: 10.1044/jshd.3204.336. No abstract available. PMID 6074893
- [Background] Dalzell L, Orlando M, MacDonald M, Berg A, Bradley M, Cacace A, Campbell D, DeCristofaro J, Gravel J, Greenberg E, Gross S, Pinheiro J, Regan J, Spivak L, Stevens F, Prieve B. The New York State universal newborn hearing screening demonstration project: ages of hearing loss identification, hearing aid fitting, and enrollment in early intervention. Ear Hear. 2000 Apr;21(2):118-30. doi: 10.1097/00003446-200004000-00006. PMID 10777019
- [Background] Chapman DA, Stampfel CC, Bodurtha JN, Dodson KM, Pandya A, Lynch KB, Kirby RS. Impact of co-occurring birth defects on the timing of newborn hearing screening and diagnosis. Am J Audiol. 2011 Dec;20(2):132-9. doi: 10.1044/1059-0889(2011/10-0049). Epub 2011 Sep 22. PMID 21940980
- [Background] Byl FM Jr. Sudden hearing loss: eight years' experience and suggested prognostic table. Laryngoscope. 1984 May;94(5 Pt 1):647-61. PMID 6325838
- [Background] Arndt S, Aschendorff A, Laszig R, Beck R, Schild C, Kroeger S, Ihorst G, Wesarg T. Comparison of pseudobinaural hearing to real binaural hearing rehabilitation after cochlear implantation in patients with unilateral deafness and tinnitus. Otol Neurotol. 2011 Jan;32(1):39-47. doi: 10.1097/MAO.0b013e3181fcf271. PMID 21068690
- [Background] Firszt JB, Holden LK, Reeder RM, Waltzman SB, Arndt S. Auditory abilities after cochlear implantation in adults with unilateral deafness: a pilot study. Otol Neurotol. 2012 Oct;33(8):1339-46. doi: 10.1097/MAO.0b013e318268d52d. PMID 22935813
- [Background] Hassepass F, Aschendorff A, Wesarg T, Kroger S, Laszig R, Beck RL, Schild C, Arndt S. Unilateral deafness in children: audiologic and subjective assessment of hearing ability after cochlear implantation. Otol Neurotol. 2013 Jan;34(1):53-60. doi: 10.1097/MAO.0b013e31827850f0. PMID 23202150
- [Background] Bishop CE, Eby TL. The current status of audiologic rehabilitation for profound unilateral sensorineural hearing loss. Laryngoscope. 2010 Mar;120(3):552-6. doi: 10.1002/lary.20735. PMID 20014322
- [Background] Essink-Bot ML, Stouthard ME, Bonsel GJ. Generalizability of valuations on health states collected with the EuroQolc-questionnaire. Health Econ. 1993 Oct;2(3):237-46. doi: 10.1002/hec.4730020307. PMID 8275169
- [Background] Chevalier J, de Pouvourville G. Valuing EQ-5D using time trade-off in France. Eur J Health Econ. 2013 Feb;14(1):57-66. doi: 10.1007/s10198-011-0351-x. Epub 2011 Sep 21. PMID 21935715
- [Background] Gaylor JM, Raman G, Chung M, Lee J, Rao M, Lau J, Poe DS. Cochlear implantation in adults: a systematic review and meta-analysis. JAMA Otolaryngol Head Neck Surg. 2013 Mar;139(3):265-72. doi: 10.1001/jamaoto.2013.1744. PMID 23429927
- [Background] Drummond M, O' brien B, Stodart G et al. 1998. Méthodes d'évaluation économique des programmes de santé. Paris : Economica, 1998.
- [Result] Marx M, Costa N, Lepage B, Taoui S, Molinier L, Deguine O, Fraysse B. Cochlear implantation as a treatment for single-sided deafness and asymmetric hearing loss: a randomized controlled evaluation of cost-utility. BMC Ear Nose Throat Disord. 2019 Feb 4;19:1. doi: 10.1186/s12901-019-0066-7. eCollection 2019. PMID 30766449
- [Derived] Dorbeau C, Galvin J, Fu QJ, Legris E, Marx M, Bakhos D. Binaural Perception in Single-Sided Deaf Cochlear Implant Users with Unrestricted or Restricted Acoustic Hearing in the Non-Implanted Ear. Audiol Neurootol. 2018;23(3):187-197. doi: 10.1159/000490879. Epub 2018 Oct 23. PMID 30352440